CLINICAL TRIAL: NCT03900806
Title: Internet-based WOrk-related Cognitive Rehabilitation for Cancer Survivors: a Randomized Controlled Trial
Acronym: i-WORC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other); Amsterdam UMC, location VUmc (Other); Maastricht University Medical Center (Other); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M18IWO
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Problems
Keywords: Cancer, Cognitive rehabilitation, eHealth
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A multicenter, three-armed randomized controlled trial will be conducted to evaluate the effectiveness of an online cognitive rehabilitation program. Two intervention groups (i.e., an extensive and a basic cognitive rehabilitation program) and one waitlist control group will be included. An economic evaluation will be conducted to assess cost-effectiveness of the cognitive rehabilitation program.
Masking Description: Blinding of participants and professionals is not possible for this type of intervention. Blinding for assessment is not applicable since measurements are computer-based.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic Cognitive Rehabilitation (Experimental): The basic arm will consist of a brief cognitive training programme without individual guidance throughout the intervention, involving three to five sessions (each approximately 60 minutes in duration), which have to be completed in a period of 12 weeks.
  Interventions: Behavioral: online cognitive rehabilitation
- Extensive Cognitive Rehabilitation (Experimental): The extensive arm will consist of a comprehensive training program, involving five to eight sessions (each approximately 60 minutes in duration), which have to be completed in a period of 12 weeks. After the first session, each further session in the extensive group involves tailored therapy guidance . Cognitive strategy modules will be assigned by the therapist depending on the participants' cognitive profile and personal treatment goals.
  Interventions: Behavioral: online cognitive rehabilitation
- Waitlist control group (No Intervention): Participants in the waiting list control group will be offered the opportunity to follow the basic cognitive rehabilitation program after completion of the 26-week follow-up measurement.

INTERVENTIONS:
Behavioral: online cognitive rehabilitation — The cognitive rehabilitation program will be based on the protocol of a frequently used meta-cognitive strategy approach applied in many rehabilitation centers in the Netherlands. The program consists of several modules that can be used in a flexible way, depending on the specific individual problems and goals. Therapists have undergone additional training in issues related to cancer-related cognitive impairment and problems occupationally active cancer survivors might experience at work. In both intervention arms, participants will receive access to a secured personal webpage, where all content relevant to the treatment sessions can be obtained.
  Arms: Basic Cognitive Rehabilitation; Extensive Cognitive Rehabilitation

SUMMARY:
Many of the occupationally active cancer survivors experience cognitive problems.Both from an individual and a societal perspective, it is important to sustain cancer survivors' employability.The aim of the current study is to develop an internet-based cognitive intervention programme for occupationally active cancer survivors confronted with cognitive problems, and to evaluate the (cost-)effectiveness of this program. A three-armed randomized controlled trial will be conducted with six months of follow-up, including two intervention groups (i.e., basic and extensive cognitive rehabilitation program) and one waitlist control group. Primary and secondary outcomes will be measured at baseline (T0), at three months, upon completion of the intervention (T1), and at three months post-intervention (T2).In total, 261 cancer survivors (18 - 65 years) who have returned to work and who experience cognitive problems will be recruited.

DETAILED DESCRIPTION:
The proposed study will evaluate the (cost-)effectiveness of an internet-based cognitive intervention program in achieving personal work-related rehabilitation goals in occupationally active cancer survivors confronted with cognitive problems. Secondary outcomes will be among others subjective cognitive function, work function and quality of life.

It is hypothesized that:

* both cancer survivors who undergo the basic or extensive cognitive rehabilitation program will achieve better their pre-set rehabilitation goals, both at baseline till treatment endpoint (T1) and follow-up (T2), compared to cancer survivors in the waitlist control group.
* cancer survivors with baseline cognitive deficits (measured with neuropsychological tests) will achieve better their pre-set rehabilitation goals after the extended cognitive rehabilitation program than after the basic cognitive rehabilitation program.

A three-armed randomized controlled trial with two intervention groups (i.e., an extensive and a basic cognitive rehabilitation program) and one waitlist control group will be conducted.

The cognitive rehabilitation program will be delivered online; either as a self-help intervention or as an online therapist-guided intervention. The therapists will be cognitive trainers who have undergone additional training in issues related to cancer-related cognitive decline.

Participants will be followed for six months in total, including three measurements time points (at baseline (T0), at three months (treatment endpoint; T1) and at 6 months follow-up (three months after completion of treatment; T2).

Cancer patients will be identified through the tumour registry, in case of the Netherlands Cancer Institute, or through the Netherlands Cancer Registry (IKNL), in all other centers. Patients will be recruited via their treating physician using an information letter of the study, including a response card. If patients are interested in participation, a member of the study team will call the patient to provide them with further information and to screen for eligibility.

Sample size calculation: This longitudinal study design will allow for testing of the main effect of the intervention (exposure to a cognitive rehabilitation programme) over time, with the GAS score as the primary outcome measure. With a sample size of 65, and alpha =0.05, the study will allow for an attrition rate of approximately 20% and have 80% power to detect an effect size of f=0.2 (equivalent to Cohens d =0.4) for the main effect of the intervention between both the basic- and extended cognitive rehabilitation treatment group and the waitlist control group. To perform subgroup analysis, as indicated by our second aim, sample size should be inflated fourfold. Therefore, we strive for a sample size of 261, with 87 patients in each group.

The intervention arms differ with respect to therapy guidance and intensity of the cognitive rehabilitation part. Both programs involve psychoeducation, cognitive behavioural therapy and fatigue management. In both intervention arms, participants will receive access to a secured personal webpage where all content relevant to the treatment sessions can be obtained.

Prior to randomization, a face-to-face appointment with a therapist will be convened to discuss the results of the neuropsychological tests, to evaluate the self-perceived (cognitive) complaints and to define three primary work-related intervention goals.

Upon receipt of all baseline information and one face-to-face session with a cognitive therapist (involving feedback on baseline neuropsychological tests and personalized treatment goal setting) , patients will be randomly allocated to the basic arm (N=87), the extensive arm (N = 87) or the waitlist control group (N = 87), using the computerized randomization programme ALEA. Stratified randomization will be applied for cognitive impairment on tests (yes/no). Minimization will be applied with respect to cognitive impairment status to equalize group sizes. Blinding of participants and professionals is not possible for this type of intervention. Blinding for assessment is not applicable since measurements are computer-based.

Study procedures: All eligible patients will be asked to complete an online neuropsychological assessment and patient-reported outcomes regarding cognition, work-related functioning and overall health-related quality of life at baseline (T0). As noted previously, results of baseline information and subsequently intervention goals will be discussed with patients prior to randomisation. Upon completion of the intervention (T1) and at three months post-intervention (T2), primary and secondary outcomes will be assessed through online questionnaire and through a call with the cognitive therapist in case of goal attainment. Participants in the waitlist control group will be given the choice to undergo the online rehabilitation programme after T2. Finally, non-response will be measured by assessing the proportion of patients who participated in comparison with all eligible patients.

Intervention effectiveness will be measured in terms of work-related goal attainment and secondary outcome measures. Furthermore, secondary analysis will be performed to explore mediating and moderating processes.

Cost-effectiveness: An economic evaluation will be conducted alongside the randomized controlled trial to evaluate costs and patient outcomes of implementing the online cognitive rehabilitation programme. From a societal perspective, a cost-utility analysis (CUA) will be conducted, whereby all costs and consequences are taken into account irrespective of who pays or benefits from them. Furthermore, in order to sustain cost-effectiveness from an employer's point of view, we will conduct a cost-effectiveness analysis (CEA) to compare the difference in costs versus the difference in effects over the two intervention groups and the waitlist control group. The cost-effectiveness of the two interventions will be evaluated by incremental treatment costs for improving goal attainment by a clinically relevant degree.

STATISTICAL ANALYSIS Means and SDs will be presented for continuous normally distributed variables and median and regions for non-normally distributed variables.

Baseline characteristics: Analyses will first be performed to evaluate the comparability of the control and the intervention groups (basic and expanded cognitive rehabilitation) at baseline in terms of sociodemographic and clinical characteristics. ANOVA tests or appropriate non-parametric statistics will be used, depending on the level of measurement. If, despite the stratified randomization procedures, the groups are found not to be comparable on one or more background variables, those variables will be employed as covariates in subsequent analyses.

GAS will be used as the primary study endpoint, evaluating between-group differences over time in GAS-scores. The GAS scores will be calculated according to published scoring algorithms. To evaluate the intra-individual difference in the trajectory of change over time for the primary outcome, we will use a growth curve modeling approach with random intercept and slope. This approach takes into account the within and between person variability, and deals adequately with missing data. Both linear and quadratic effect of time will be modeled to determine if an initial improvement or deterioration in the outcome was followed by a deceleration of this change over time. Appropriateness of the final model (with or without quadratic effect) will be determined based on model fit statistics: the Bayesian information criterion (BIC; Schwarz, 1978) and the Akaike information criterion (AIC; Akaike, 1998). In all analyses the control group will be the reference group. Furthermore, moderation analysis will be conducted to determine whether the interventions have a differential effect among the subgroups classified as cognitive impaired yes or no (measured by ACS) at baseline. The same approach will be used for secondary outcome measures.

All analyses will be done on an ´intention to treat´ basis. Differences in mean change scores over time between the intervention groups and the control group will be accompanied by effect sizes.

ELIGIBILITY:
Inclusion Criteria:

1. Working age (18 - 65 years) at the time of study entry
2. Histologically confirmed cancer (all tumour types except for brain tumours).
3. Completed primary therapy including chemotherapy, targeted agents and/or immunotherapy 6 months ago. Patients who are still receiving hormonal therapy can be included in the trial.
4. Experience cancer/cancer treatment-related cognitive problems. Both patients with and without cognitive impairment assessed with neuropsychological tests, formally assessed with neuropsychological tests, will be included in the study.
5. Fixed or temporary employment contract (with at least six months left of their contract).
6. Being at work for a minimum of 12 working hours/week.

Exclusion Criteria:

1. Psychiatric or neurological disorder that can interfere with current study aims.
2. Lack basic proficiency in Dutch.
3. Participating in comparable studies or programmes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2019-08-03 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Goal Attainment Scaling (GAS) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Individually defined work-related treatment goals will be measured using the 6-point Goal Attainment Scale (GAS) on personal outcome (-3, achievement of the goal after training is worse; -2, achievement of the goal is the same; 1, partial achievement of the goal; 0, achievement of the goal; 1, exceeding the goal, and 2, greatly exceeding the goal). Patients will formulate three treatment goals at baseline, in collaboration with their cognitive therapist. Attainment of the goals is measured in a standardized way, i.e., an overall GAS T-score will be computed for each participant on basis of aggregated GAS scores involving attainment of multiple personal treatment goals, according a summary scoring algorithm that calculates the extent to which patients' goals are met.

SECONDARY OUTCOMES:
Change from baseline Cognitive problems (CSC-W DV) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Self-perceived cognitive problems will be assessed using the Cognitive Symptom Checklist-Work, Dutch version (CSC-W DV). This 19-item questionnaire for measuring work-related cognitive problems in cancer patients contains an ordinal five-point scale, ranging from 0 (never) to 4 (always). An additional response option 'does not apply to my job' is used in case a particular symptom is not relevant to the participants job. Total scores will be obtained by summing the scores on each item, divided by the number of items and then multiplied by 25 to obtain scores between 0 and 100, with higher scores indicating more cognitive symptoms. The scores on 'does not apply to my job' will be transformed to missing values.
Change from baseline Work ability (WAI) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Work ability will be assessed using the first item of the Work Ability Index (WAI), asking participants to estimate their current work ability compared to their lifetime best (0, cannot work at all, to 10, best ever). This first overall single item correlates correlates with the total work ability score.
Change from baseline Work functioning (WRFQ) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Work functioning among participants will be measured using the 27-item Work Role Functioning Questionnaire (WRFQ), distinguishing five different work domains: work scheduling demands, mental demands, social demands, physical demands, and output demands (range 0 to 100). Higher scores indicate better work functioning.
Change from baseline Need for recovery after a work day (VBBA) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Need for recovery after a workday will be assessed using the dichotomous (yes/no) 11-item subscale of the questionnaire on Perception and Judgement of Work (VBBA). Examples of this items are: "I find it difficult to relax after a working day" and "When I come home from work people should leave me alone".
Change in Health-Related Quality of Life (SF-36) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Health-Related Quality of Life will be measured using the SF-36. This 36-item list consists of eight functional scales (i.e., vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, mental health, emotional role functioning, and social role functioning).
Change from baseline Fatigue (SF-36) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Fatigue will be measured with the subscale vitality of the SF-36, as this shows to be a valid measure of cancer-related fatigue.
Change from baseline Neuropsychological functioning (ACS) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Neuropsychological functioning will be measured using a self-administered online neuropsychological test battery, the Amsterdam Cognition Scan (ACS). The ACS distinguishes the following cognitive domains: executive functioning, information processing speed, attention, working memory, verbal learning and memory, processing speed, psychomotor speed. In total, the ACS consists out of seven different neuropsychological tasks. Participants are asked to complete the test in one setting of approximately 75 minutes, in which two fixed breaks for 2 minutes are included. The ASC is usable a reliable for the oncology setting, with test-retest correlations in the range 0.29 up to 0.78, which is comparable with traditional tests. Furthermore, concurrent validity with traditional tests is medium to large.
Change from baseline Job characteristics (JCQ) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Job characteristics will be measured with the Dutch version of the Job Content Questionnaire (JCQ). Five different domains of job characteristics will be assessed, namely decision latitude (composite score of the subscales skill discretion and decision authority), psychological demands, physical job demands, job insecurity and social support (composite score of subscales supervisor social support, and co-worker social support). In total, this will result in 35 items with ordinal four-point scales, ranging from 1 (totally disagree) to 4 (totally agree).
Change from baseline Coping (CERQ) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Coping will be assessed with the 5-point Cognitive Emotion Regulation Questionnaire (CERQ), involving 36 items measuring 9 different coping styles (i.e. self-blame, acceptance, rumination, positive refocusing, refocus of planning, positive reappraisal, putting in to perspective, catastrophizing and other blame).
Change from baseline Depression and anxiety (HADS) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Depression and anxiety will be assessed with the 4-point Hospital Anxiety and Depression Scale (HADS), involving two 7-item subscales: anxiety and depression. A score of 11 and over indicates the possible presence of clinical depression.
Change from baseline Work involvement (WIS) at 3 and 6 months follow-up. | T0 (baseline), T1 (12 weeks), T2 (26 weeks)
  Work involvement (the importance of work and values about the goodness of work) will be assessed with the Work Involvement Scale (WIS), involving six items rated on a five-point scale (1 = totally disagree to 5 = totally agree). High scores indicate a high work involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Sanne B. Schagen, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klaver KM, Duijts SFA, Geusgens CAV, Kieffer JM, Agelink van Rentergem J, Hendriks MP, Nuver J, Marsman HA, Poppema BJ, Oostergo T, Doeksen A, Aarts MJB, Ponds RWHM, van der Beek AJ, Schagen SB. Internet-based cognitive rehabilitation for working cancer survivors: results of a multicenter randomized controlled trial. JNCI Cancer Spectr. 2024 Jan 4;8(1):pkad110. doi: 10.1093/jncics/pkad110. PMID 38273712
- [Derived] Klaver KM, Duijts SFA, Geusgens CAV, Aarts MJB, Ponds RWHM, van der Beek AJ, Schagen SB. Neuropsychological test performance and self-reported cognitive functioning associated with work-related outcomes in occupationally active cancer survivors with cognitive complaints. J Cancer Surviv. 2024 Apr;18(2):412-424. doi: 10.1007/s11764-022-01223-x. Epub 2022 Jul 1. PMID 35776235
- [Derived] Klaver KM, Duijts SFA, Geusgens CAV, Aarts MJB, Ponds RWHM, van der Beek AJ, Schagen SB. Internet-based cognitive rehabilitation for WORking Cancer survivors (i-WORC): study protocol of a randomized controlled trial. Trials. 2020 Jul 20;21(1):664. doi: 10.1186/s13063-020-04570-1. PMID 32690067